CLINICAL TRIAL: NCT05803473
Title: In-hospital Diabetes Management by a Diabetes Team and Continuous Glucose Monitoring or Point of Care Glucose Testing (DIATEC): a Randomised Trial
Brief Title: DIAbetes TEam and Cgm in Managing Hospitalised Patients with Diabetes
Acronym: DIATEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Kristensen (Other)
Responsible Party: Sponsor-Investigator, Peter Kristensen, Medical Doctor, PhD, Clinical Associate Professor, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2301240
Record Dates: First submitted 2023-03-14; First posted 2023-04-07 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Inpatient; Randomised controlled trial; Hyperglycemia; Hypoglycemia; Glycemic variabiity; Continuous glucose monitoring; CGM; In-hospital; Telemetric continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, two-site, prospective randomised open-label blinded endpoint (PROBE) trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- POC-arm (Active Comparator): Subjects are monitored by point-of-care (POC) glucose testing. Diabetes management is done by usual ward nurses and guided by an in-hospital diabetes team. A blinded CGM is mounted in the POC-arm for outcome analysis.
  Interventions: Device: FreeStyle Precision Pro Glucometer for glucose POC testing
- CGM-arm (Experimental): CGM-arm subjects are monitored by CGM viewed by the in-hospital diabetes team in addition to POC glucose testing performed by usual ward nurses. Diabetes management is done by usual ward nurses by POC glucose testing and guided by an in-hospital diabetes team with acces to CGM data.
  Interventions: Device: Dexcom G6 Continuous Glucose Monitoring System (Dexcom Inc., San Diego, USA)

INTERVENTIONS:
Device: Dexcom G6 Continuous Glucose Monitoring System (Dexcom Inc., San Diego, USA) — For CGM-arm subjects, glucose data are obtained by the CGM Dexcom G6 which via an iPhone SE 3 transmits data to the in-hospital diabetes team stations to be displayed on an iPad 9 10.2".
  Arms: CGM-arm
Device: FreeStyle Precision Pro Glucometer for glucose POC testing — For the POC-arm subjects, glucose assessment is done by standard ward glucometer.
  Arms: POC-arm

SUMMARY:
This trial investigates the effects of continuous glucose monitoring (CGM) and an in-hospital diabetes team on in-hospital glycemic and clinical outcomes in patients with type 2 diabetes compared to standard glucose point-of-care (POC) testing and an in-hospital diabetes team.

DETAILED DESCRIPTION:
In Denmark and worldwide, 15-20 % of hospitalised patients have diabetes mellitus. For most patients, diabetes is not the primary cause of admission. The patients are therefore under the care of non-diabetes specialists. Consequently, diabetes management can be inadequate resulting in hypoglycemia, hyperglycemia, and increased glycemic variability, which might increase patient mortality, morbidity, and length of hospital stay. Despite these challenges, a recent review concludes that in-hospital diabetes management is under-researched. Therefore, new in-hospital diabetes management strategies are greatly needed.

Continuous glucose monitoring (CGM) might accommodate this need by providing 288 glucose readings per day compared to usual glucose point-of-care (POC) testing from finger-prick blood 3-5 times per day during admission. CGM glucose levels can be transmitted from the patient's room to a monitoring screen at the nursing stations. This setup is called telemetric CGM. Outstanding results on glycemic and clinical outcomes in an out-hospital setting exist, however, In-hospital CGM has been associated only with a clinically insignificant reduction of mean daily glucose levels and a small increased detection rate of hypoglycemia of glucose levels <3 mmol/L (<54 mg/dL) compared to POC. Reasons for this might be that an in-hospital diabetes team (i.e., educated diabetes nurses with CGM competencies) is imperative in achieving optimal use of telemetric CGM.

This trial investigates if telemetric CGM and an in-hospital diabetes team improve patients' in-hospital glycemic and clinical outcomes compared to POC glucose testing and an in-hospital diabetes team

ELIGIBILITY:
Inclusion Criteria:

* A documented history of T2DM prior to inclusion
* Age ≥ 18 years old
* Willingness and ability to comply with the clinical investigation plan
* Ability to communicate in Danish with the trial personnel
* An expected length of hospital stay for at least two days after enrolment
* If subject with childbearing potential (subject < 50 years old); willing to have a urine pregnancy test performed and/or to use a highly effective method of contraception (i.e., birth control implant, intrauterine device, birth control shot, or sterilisation).

Exclusion Criteria:

* Patients on out-hospital basal insulin with duration of action > 24 hours (Toujeo or Tresiba)
* Treated with hydroxyurea/hydroxycarbamid
* Nutritional therapy (continuous enteral or parenteral feeding)
* Clinically relevant pancreatic disease
* Systemic glucocorticoid treatment with prednisone equivalent dose >5 mg/day
* Expected to require admission to the intensive-care unit
* Anasarca (severe and general edema)
* Dialysis
* Estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m2
* Known hypersensitivity to the band-aid of the CGM Dexcom G6 sensor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Time in range | During hospitalization (up to 30 days)
  Time in range (TIR) is defined as the percentage of time within glucose level of 3.9-10.0 mmol/L (70-180 mg/dL) measured by CGM.

SECONDARY OUTCOMES:
Time in range per day 3.9-10.0 mmol/L (70-180 mg/dL) | During hospitalization (up to 30 days)
  Percentage of time in range assessed each day of inclusion; amount of time (hours and minutes).
Time above range (TAR) >10.0 mmol/L (>180 mg/dL) | During hospitalization (up to 30 days)
  Percentage of time above range; amount of time (hours and minutes).
Time above range (TAR) >13.9 mmol/L (>250 mg/dL) | During hospitalization (up to 30 days)
  Percentage of time above range; amount of time (hours and minutes).
Time below range (TBR) <3.9 mmol/L (<70 mg/dL) | During hospitalization (up to 30 days)
  Percentage of time below range; amount of time (hours and minutes)
Time below range (TBR) <3.0 (<54 mg/dL) | During hospitalization (up to 30 days)
  Percentage of time below range; amount of time (hours and minutes)
Standard deviation (SD) of all CGM glucose levels | During hospitalization (up to 30 days)
  mmol/L (mg/dL)
Coefficient of variation (CV) | During hospitalization (up to 30 days)
  SD divided by mean glucose level
Mean glucose levels | During hospitalization (up to 30 days)
  mmol/L (mg/dL)
Hypoglycemia < 3.9 mmol/L (< 70 mg/dL) | During hospitalization (up to 30 days)
  mmol/L (mg/dL), duration ≥15 consecutive min.
Hypoglycemia (level 1) 3.0-3.8 mmol/L (54-69 mg/dL) | During hospitalization (up to 30 days)
  mmol/L (mg/dL), duration ≥15 consecutive min.
Hypoglycemia (level 2) < 3.0 mmol/L (<54 mg/dL) | During hospitalization (up to 30 days)
  mmol/L (mg/dL), duration ≥15 consecutive min.
Recurrent hypoglycemic events | During hospitalization (up to 30 days)
  Number; Reoccurring hypoglycemic events after the first episode of hypoglycemia.

OTHER OUTCOMES:
Length of hospital stay | During hospitalization (up to 30 days)
  The length of hospital stay from inclusion to discharge.
Number of In-hospital complications | During hospitalization (up to 30 days)
  Any in-hospital related complications occurring at least one day after randomisation (e.g. acute kidney injury, death during hospitalisation, transfer to intensive care unit etc.).
Number of times insulin is administered | During hospitalization (up to 30 days)
  The number of times basal, prandial, and correctional insulin is used in total and correctly used according to clinical investigation plan specifications.
Insulin doses | During hospitalization (up to 30 days)
  Basal, prandial, and correctional insulin doses in total.
Readmissions and mortality | 30-day after discharge from hospital
  Assesment of 30-day numbers of readmissions and mortality.
Questionnaires | During hospitalization (up to 30 days)
  Subject and in-hospital diabetes team user satisfaction levels with in-hospital telemetric CGM are assessed by validated questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lommer Kristensen, MD, PhD, Principal Investigator — Copenhagen University Hospital - North Zealand, Department of Endocrinology and Nephrology, Denmark; Katrine Bagge Hansen, MD, PhD, Principal Investigator — Copenhagen University Hospital - Herlev-Gentofte, Steno Diabetes Center Copenhagen, Denmark
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital - Herlev-Gentofte (Steno Diabetes Center Copenhagen), Herlev
  - Copenhagen University Hospital - North Zealand, Hillerød

IPD SHARING:
Plan to Share IPD: Yes
If required by medical journal to which articles are planned to be submitted or by request to corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available at the end of the trial. Anticipation: Year 2025
Access Criteria: Supporting information is available by request to corresponding author of the planned articles when the trial is completed.

REFERENCES:
- [Background] Umpierrez GE, Isaacs SD, Bazargan N, You X, Thaler LM, Kitabchi AE. Hyperglycemia: an independent marker of in-hospital mortality in patients with undiagnosed diabetes. J Clin Endocrinol Metab. 2002 Mar;87(3):978-82. doi: 10.1210/jcem.87.3.8341. PMID 11889147
- [Background] Kristensen PL, Jessen A, Houe SMM, Banck-Petersen P, Schiotz C, Hansen KB, Svendsen OL, Almdal T, Bjerre-Christensen U. Quality of diabetes treatment in four orthopaedic departments in the Capital Region of Denmark. Dan Med J. 2021 Nov 30;68(12):A05210449. PMID 34851255
- [Background] Akiboye F, Sihre HK, Al Mulhem M, Rayman G, Nirantharakumar K, Adderley NJ. Impact of diabetes specialist nurses on inpatient care: A systematic review. Diabet Med. 2021 Sep;38(9):e14573. doi: 10.1111/dme.14573. Epub 2021 May 18. PMID 33783872
- [Background] Swanson CM, Potter DJ, Kongable GL, Cook CB. Update on inpatient glycemic control in hospitals in the United States. Endocr Pract. 2011 Nov-Dec;17(6):853-61. doi: 10.4158/EP11042.OR. PMID 21550947
- [Background] Thabit H, Hovorka R. Glucose control in non-critically ill inpatients with diabetes: towards closed-loop. Diabetes Obes Metab. 2014 Jun;16(6):500-9. doi: 10.1111/dom.12228. Epub 2013 Nov 24. PMID 24267153
- [Background] Olsen MT, Dungu AM, Klarskov CK, Jensen AK, Lindegaard B, Kristensen PL. Glycemic variability assessed by continuous glucose monitoring in hospitalized patients with community-acquired pneumonia. BMC Pulm Med. 2022 Mar 9;22(1):83. doi: 10.1186/s12890-022-01874-7. PMID 35264139
- [Background] Baker EH, Janaway CH, Philips BJ, Brennan AL, Baines DL, Wood DM, Jones PW. Hyperglycaemia is associated with poor outcomes in patients admitted to hospital with acute exacerbations of chronic obstructive pulmonary disease. Thorax. 2006 Apr;61(4):284-9. doi: 10.1136/thx.2005.051029. Epub 2006 Jan 31. PMID 16449265
- [Background] Dhatariya KK, Umpierrez G. Gaps in our knowledge of managing inpatient dysglycaemia and diabetes in non-critically ill adults: A call for further research. Diabet Med. 2023 Mar;40(3):e14980. doi: 10.1111/dme.14980. Epub 2022 Nov 16. PMID 36256494
- [Background] Klarskov CK, Windum NA, Olsen MT, Dungu AM, Jensen AK, Lindegaard B, Pedersen-Bjergaard U, Kristensen PL. Telemetric Continuous Glucose Monitoring During the COVID-19 Pandemic in Isolated Hospitalized Patients in Denmark: A Randomized Controlled Exploratory Trial. Diabetes Technol Ther. 2022 Feb;24(2):102-112. doi: 10.1089/dia.2021.0291. Epub 2022 Jan 4. PMID 34524009
- [Background] Seisa MO, Saadi S, Nayfeh T, Muthusamy K, Shah SH, Firwana M, Hasan B, Jawaid T, Abd-Rabu R, Korytkowski MT, Muniyappa R, Antinori-Lent K, Donihi AC, Drincic AT, Luger A, Torres Roldan VD, Urtecho M, Wang Z, Murad MH. A Systematic Review Supporting the Endocrine Society Clinical Practice Guideline for the Management of Hyperglycemia in Adults Hospitalized for Noncritical Illness or Undergoing Elective Surgical Procedures. J Clin Endocrinol Metab. 2022 Jul 14;107(8):2139-2147. doi: 10.1210/clinem/dgac277. PMID 35690929
- [Derived] Olsen MT, Klarskov CK, Pedersen-Bjergaard U, Hansen KB, Kristensen PL. Summary of clinical investigation plan for The DIATEC trial: in-hospital diabetes management by a diabetes team and continuous glucose monitoring or point of care glucose testing - a randomised controlled trial. BMC Endocr Disord. 2024 May 6;24(1):60. doi: 10.1186/s12902-024-01595-4. PMID 38711112